CLINICAL TRIAL: NCT03200301
Title: Effect of Intact Umbilical Cord Milking Versus Immediate Cord Clamping on Neonatal Outcomes and First Year Neurodevelopmental Outcomes in Very Preterm Infants - A Randomised Controlled Trial
Brief Title: Effect of Intact Umbilical Cord Milking on Neonatal and First Year Neurodevelopmental Outcomes in Very Preterm Infants.
Acronym: Cord-milking
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Jubilee MMCRI
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Preterm Infant; Umbilical Cord Milking
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intact Umbilical Cord Milking (Experimental): Umbilical Cord Milking involves pinching of the cord close to the placenta and milking about 20 cm segment of the cord proximal to the umbilicus, towards the infant over a 2-second duration. The cord will be then released, allowing for a brief 2-second pause between each milking motion. This will be repeated for a total of 3 times over a duration less than 20 seconds.
  Interventions: Procedure: Intact Umbilical Cord Milking
- Early Cord Clamping (No Intervention): Umbilical cord will be clamped immediately after delivery and baby will be handed over to the neonatal team.

INTERVENTIONS:
Procedure: Intact Umbilical Cord Milking — Immediately after delivery, the infant will be placed at or ∼20 cm below the level of the placenta and about 20 cm of the intact umbilical cord will be milked towards the umbilicus three times. The technique consists of pinching the cord close to the placenta and milking about 20 cm segment of the cord proximal to the umbilicus, towards the infant over a 2-second duration. The cord will then be released and allowed to refill with blood for a brief 2-second pause between each milking motion. After completion of milking three times, the cord will be clamped close to the umbilicus and the neonate handed over to the neonatal team. The procedure of cord milking will be completed within 20 seconds.
  Other Names: Milking of the Umbilical Cord
  Arms: Intact Umbilical Cord Milking

SUMMARY:
The investigators hypothesise that intact umbilical cord milking (I-UCM) will reduce neonatal morbidity and improve long term neurodevelopmental outcome in very preterm infants. All babies born less than 32 weeks gestation, meeting the inclusion criteria will be randomly assigned to either I-UCM or immediate cord clamping (ICC) and their short and long term outcome measures analyzed.

DETAILED DESCRIPTION:
Optimizing placental transfusion at birth promotes a more physiologic transition from intrauterine to extrauterine life. There is increasing evidence about the benefits of enhanced placental transfusion in improving neonatal outcomes, such as higher hemoglobin concentration, improved hemodynamic stability, reduced incidence of intraventricular hemorrhage, less need for blood transfusions and better neurodevelopmental outcome in preterm infants.

The investigators propose to evaluate the the safety and effectiveness of I-UCM versus ICC in mothers undergoing preterm delivery before 32 weeks, by randomly assigning them to one of two groups - study and control. The study group will undergo I-UCM during delivery and the control group will have ICC, which is the current standard of care. Both groups will subsequently receive routine care for mother and infant. In the study group the infants will be placed at or ∼20 cm below the level of the placenta and about 20 cm of the intact umbilical cord will be milked towards the umbilicus three times. The technique consists of pinching the cord close to the placenta and milking about 20 cm segment of the cord proximal to the umbilicus, towards the infant over a 2-second duration. The cord will then be released and allowed to refill with blood for a brief 2-second pause between each milking motion. After completion of milking three times, the cord will be clamped close to the umbilicus and the neonate handed over to the neonatal team. The procedure of cord milking will be completed within 20 seconds.

Prenatal and delivery data will be collected from the mother's charts. Infant data will be collected from hospital admission records and from follow up for a period up to 12 months of corrected age. The infant data collected will include hemoglobin levels at birth, incidence and severity of intraventricular hemorrhage in the first week of life and neonatal morbidity (resuscitation measures, peak bilirubin, need for phototherapy and blood transfusion, sepsis, necrotizing enterocolitis, retinopathy of prematurity and chronic lung disease) and mortality. The neurodevelopmental status of both the study and control group of infants will be assessed at 6 months and one year of corrected age. The investigators hypothesize that I-UCM provides a greater placental transfusion and better neonatal outcomes when compared to ICC. It is a simple procedure which can be practiced universally and of great relevance to both developed and developing countries.

ELIGIBILITY:
Inclusion Criteria:

* All the preterm infants of less than 32 weeks of gestation born of consenting parents in the hospital

Exclusion Criteria:

* Neonates depressed at birth, MCMA, MCDA Twin pregnancy (DCDA twins are included), Severe IUGR in antenatal scans (< 10th Centile), Known case of Hydrops fetalis, Known major congenital anomaly, Placenta previa and abruptions, bleeding, accreta, nuchal cord, anhydramnios, PROM > 2 weeks before 24 weeks and Refusal to Consent by the Parents

Ages: 1 Minute to 5 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Haemoglobin levels at birth | 1 hour
  Haemoglobin levels at birth
Intraventricular Haemorrhage | 7 days of life
  Incidence and severity of Intraventricular Haemorrhage in the first week of life - Cranial Ultrasound done on day 7

SECONDARY OUTCOMES:
The resuscitation interventions required with and without umbilical cord milking. | 20 minutes after delivery
  The resuscitation interventions required that will be assessed are requirement of Continuous Positive Airway Pressure (CPAP), oxygen, mask and bag ventilation, endotracheal intubation and ventilation, chest compressions, drugs, and fluid boluses
Resuscitation outcomes with and without umbilical cord milking. | 20 minutes after delivery
  Short term outcomes of resuscitation will be assessed using the validated Combined Apgar score (consisting of the Expanded and Specified Apgar scoring systems) introduced by Rudiger et al, in depressed neonates with and without UCM.
  Ref:Dalili H, Nili F, Sheikh M, Hardani AK, Shariat M, Nayeri F (2015) Comparison of the Four Proposed Apgar Scoring Systems in the Assessment of Birth Asphyxia and Adverse Early Neurologic Outcomes. PLoS ONE 10(3): e0122116
Incidence of hypotension | 24 hours of life
  Incidence of hypotension
Requirement of inotropic support | 24 hours of life
  Number of inotropes required for support
symptomatic polycythemia | 48 hours of life
  The number of neonates with symptomatic polycythemia (defined as lethargy, plethora, jitteriness, tachycardia, tachypnea and with venous hematocrit > 65%).
Sepsis (culture positive) | 72 hours of life
  Incidence of Sepsis (culture positive)
Peak bilirubin levels | 72 hours of life
  Serum peak bilirubin levels
Requirement of phototherapy or exchange transfusion | 72 hours of life
  Neonates requiring phototherapy or exchange transfusion will be evaluated according to the NICE guidelines and serum bilirubin levels will be interpreted according to the baby's age in hours. Physicians who assess the neonate and advice phototherapy or exchange transfusion will be blinded to the intervention.
Incidence of Necrotising Enterocolitis (NEC) | 14 days of life
  Incidence of Necrotising Enterocolitis as defined by modified Bell's Criteria
Requirement of Oxygen | 36 weeks of gestational age
  Requirement of Oxygen at 28 days of life and at 36 weeks gestation
Requirement of red blood cell transfusions | 4 weeks of life
  Requirement of red blood cell transfusions before discharge
Number of days of Hospital Stay after Birth | 4 weeks of life
  Number of days of Hospital Stay after Birth
Death prior to discharge | 4 weeks of life
  Death prior to discharge
Serum iron stores | 6 months of age
  Serum iron stores (ferritin levels) at 6 weeks and 6 months of age
Developmental Assessment Scales for Indian Infants (DASII) | 1 year of corrected age
  Developmental Assessment Scales for Indian Infants (DASII) tests carried out at 6 months and 1 year of corrected age. The DASII scale is divided into motor scale and mental scale. The motor scale consists of 67 items and mental scale consists of 163 items. (P Phatak, et al, 1996)

CONTACTS AND LOCATIONS:
Locations (1):
- Jubilee Mission Medical College & Research Institute, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Wassia H, Shah PS. Efficacy and safety of umbilical cord milking at birth: a systematic review and meta-analysis. JAMA Pediatr. 2015 Jan;169(1):18-25. doi: 10.1001/jamapediatrics.2014.1906. PMID 25365246
- [Background] Boere I, Roest AA, Wallace E, Ten Harkel AD, Haak MC, Morley CJ, Hooper SB, te Pas AB. Umbilical blood flow patterns directly after birth before delayed cord clamping. Arch Dis Child Fetal Neonatal Ed. 2015 Mar;100(2):F121-5. doi: 10.1136/archdischild-2014-307144. Epub 2014 Nov 11. PMID 25389141
- [Background] Katheria AC, Brown MK, Rich W, Arnell K. Providing a Placental Transfusion in Newborns Who Need Resuscitation. Front Pediatr. 2017 Jan 25;5:1. doi: 10.3389/fped.2017.00001. eCollection 2017. PMID 28180126
- [Background] Katheria AC, Truong G, Cousins L, Oshiro B, Finer NN. Umbilical Cord Milking Versus Delayed Cord Clamping in Preterm Infants. Pediatrics. 2015 Jul;136(1):61-9. doi: 10.1542/peds.2015-0368. PMID 26122803
- [Background] Rabe H, Sawyer A, Amess P, Ayers S; Brighton Perinatal Study Group. Neurodevelopmental Outcomes at 2 and 3.5 Years for Very Preterm Babies Enrolled in a Randomized Trial of Milking the Umbilical Cord versus Delayed Cord Clamping. Neonatology. 2016;109(2):113-9. doi: 10.1159/000441891. Epub 2015 Dec 10. PMID 26650133
- [Background] Ghavam S, Batra D, Mercer J, Kugelman A, Hosono S, Oh W, Rabe H, Kirpalani H. Effects of placental transfusion in extremely low birthweight infants: meta-analysis of long- and short-term outcomes. Transfusion. 2014 Apr;54(4):1192-8. doi: 10.1111/trf.12469. PMID 24843886
- [Background] Niermeyer S. A physiologic approach to cord clamping: Clinical issues. Matern Health Neonatol Perinatol. 2015 Sep 8;1:21. doi: 10.1186/s40748-015-0022-5. eCollection 2015. PMID 27057338
- [Background] Nolan JP, Hazinski MF, Aickin R, Bhanji F, Billi JE, Callaway CW, Castren M, de Caen AR, Ferrer JM, Finn JC, Gent LM, Griffin RE, Iverson S, Lang E, Lim SH, Maconochie IK, Montgomery WH, Morley PT, Nadkarni VM, Neumar RW, Nikolaou NI, Perkins GD, Perlman JM, Singletary EM, Soar J, Travers AH, Welsford M, Wyllie J, Zideman DA. Part 1: Executive summary: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Resuscitation. 2015 Oct;95:e1-31. doi: 10.1016/j.resuscitation.2015.07.039. No abstract available. PMID 26477703
- [Background] Rabe H, Diaz-Rossello JL, Duley L, Dowswell T. Effect of timing of umbilical cord clamping and other strategies to influence placental transfusion at preterm birth on maternal and infant outcomes. Cochrane Database Syst Rev. 2012 Aug 15;(8):CD003248. doi: 10.1002/14651858.CD003248.pub3. PMID 22895933
- [Background] Safarulla A. A review of benefits of cord milking over delayed cord clamping in the preterm infant and future directions of research. J Matern Fetal Neonatal Med. 2017 Dec;30(24):2966-2973. doi: 10.1080/14767058.2016.1269319. Epub 2017 Jan 12. PMID 27936996
- [Background] Committee on Obstetric Practice, American College of Obstetricians and Gynecologists. Committee Opinion No.543: Timing of umbilical cord clamping after birth. Obstet Gynecol. 2012 Dec;120(6):1522-6. doi: 10.1097/01.AOG.0000423817.47165.48. PMID 23168790
- [Background] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001